CLINICAL TRIAL: NCT05786833
Title: Dexmedetomidine Infusion Versus Ketofol Infusion on The Incidence of Emergence Delirium in Children Undergoing Congenital Inguinal Hernia Repair: A Prospective Randomized Trial.
Brief Title: Dexmedetomidine vs Ketofol on Delirium in Children Undergoing Congenital Inguinal Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Nada Maged Shaheen, Resident of Anesthesia, Surgical Intensive Care and Pain Management ,Faculty of medicine ,Tanta University, Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 36264MS43/1/23
Record Dates: First submitted 2023-03-10; First posted 2023-03-28 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Dexmedetomidine; Ketofol; Delirium; Hernia
MeSH Terms: conditions — Delirium; Hernia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine Group (Active Comparator)
  Interventions: Drug: Dexmedetomedine
- Ketofol Group (Active Comparator)
  Interventions: Drug: Ketofol
- Control Group (Placebo Comparator)
  Interventions: Drug: isotonic saline 0.9%

INTERVENTIONS:
Drug: Dexmedetomedine — Patients will receive intraoperative dexmedetomedine intravenous infusion at a dose of 0.2µg/kg/hour.
  Arms: Dexmedetomidine Group
Drug: Ketofol — Patients will receive intraoperative ketofol (1:10 ratio of ketamine-propofol mixture) intravenous infusion with %90 of Mcfarlan dose regiment. McFarlan dose regiments include 15 mg/kg/h infusion during 15 minutes, 13 mg/kg/h infusion during second 15 minutes, 11 mg/kg/h infusion from half to 1 and 10 mg/kg/h from 1 to 2 hours.
  Arms: Ketofol Group
Drug: isotonic saline 0.9% — Patients will receive intravenous infusion of equivalent volume of isotonic saline 0.9%.
  Arms: Control Group

SUMMARY:
The aim of this study is to compare the effect of dexmedetomidine versus ketofol on the incidence of the emergence delirium in children undergoing congenital inguinal hernia repair.

DETAILED DESCRIPTION:
Emergence delirium (ED) is a disturbance in a child's awareness or attention to his/her environment with disorientation and perceptual alterations including hypersensitivity to stimuli and hyperactive motor behaviour in the immediate post anesthesia period.

Propofol is a non-opioid, non-barbiturate, sedative-hypnotic agent with rapid onset and short duration of action [12]. Ketamine is a phencyclidine derivative classified as a dissociative sedative that provides analgesia and amnesia.

Combination of ketamine with propofol reduces the sedative dose of propofol. The complementary effects of this combination are supposed to produce lower toxicity compared to each drug alone through decreasing required doses. Ketofol; mixed ketamine and propofol has been shown to be effective in emergency room for procedural sedation and for induction for rapid sequence intubation [13,14]. This combination is also effective to prevent ED in pediatric patients undergoing simple surgical procedural in addition to the advantage of better hemodynamic stability.

Dexmedetomidine is a highly selective, alpha2-adrenergic receptor agonist that has been widely used for adult anesthesia and as a sedative in intensive care units. Dexmedetomidine is safe in children due to its hypnotic, analgesic, sedative, and anxiolytic effects. it has been shown to improve intraoperative hemodynamic stability, minimize responses to stimuli, and reduce the need for other anesthetic agents.

ELIGIBILITY:
Inclusion Criteria:

* 60 children aged from 2 to 5 years
* presented with congenital inguinal hernia
* the American Society of Anaesthesiologists classification ASA I-II.

Exclusion Criteria:

* Past medical history of mental illness or neurological illness.
* Renal or hepatic diseases.
* Severe hearing or visual impairment which may interfere with communication and physical decline.
* Congenital heart disease.
* History of allergy to any of the study drugs.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-10-20 (Estimated); Study Completion 2023-10-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative emergence delirium | 5 -15 minutes
  Assessment of delirium using Pediatric Anesthesia Emergence Delirium (PAED) will be performed on arrival at the Post Anesthesia Care Unit (PACU)

CONTACTS AND LOCATIONS:
Locations (1):
- Nada Maged Shaheen, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the principal investigator
Supporting Information: Study Protocol
Time Frame: one year